CLINICAL TRIAL: NCT07216027
Title: A PHASE 2B, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, DOSE-RANGING STUDY TO EVALUATE THE EFFICACY AND SAFETY OF PF-08049820 IN ADULT PARTICIPANTS WITH MODERATE TO SEVERE ATOPIC DERMATITIS
Brief Title: A Study to Learn About Study Medicine Called PF-08049820 in People With Eczema
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C6231002; 2025-522965-31-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2025-10-09; First posted 2025-10-14 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis; Eczema, Atopic
Keywords: Eczema; Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm 1 (Experimental): Tablets taken by mouth daily for 12 weeks
  Interventions: Drug: PF-08049820
- Arm 2 (Experimental): Tablets taken by mouth daily for 12 weeks
  Interventions: Drug: PF-08049820
- Arm 3 (Experimental): Tablets taken by mouth daily for 12 weeks
  Interventions: Drug: PF-08049820
- Arm 4 (Placebo Comparator): Tablets taken by mouth daily for 12 weeks
  Interventions: Drug: Placebo
- Arm 5 (Optional) (Experimental): Tablets taken by mouth daily for 12 weeks
  Interventions: Drug: PF-08049820
- Arm 6 (Optional) (Placebo Comparator): Tablets taken by mouth daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-08049820 — Tablet
  Arms: Arm 1; Arm 2; Arm 3; Arm 5 (Optional)
Drug: Placebo — Tablet
  Arms: Arm 4; Arm 6 (Optional)

SUMMARY:
The purpose of this study is to learn if the study medicine (PF-08049820) is safe and effective for the treatment of atopic dermatitis (AD), also known as eczema, or atopic eczema. People with this condition may have severe itching and rashes on the skin.

The study is seeking participants who:

1. Are 18 years of age or more;
2. Were confirmed to have AD at least 6 months ago;
3. Do not have a suitable prescribed medicine for AD;
4. Are considered by their doctors to have moderate to severe AD.

Eligible participants will take either PF-08049820 or placebo as tablets by mouth daily for 12 weeks. A placebo does not have any medicine in it but looks just like the medicine being studied. Participants will visit the clinic on Day 1, Weeks 1, 2, 4, 6, 8 and 12, and have a follow-up visit at Week 16. During this time, the participant's health and skin condition will be checked. Participants will have blood and urine tests and must answer questions about their health, skin condition, and how much their skin condition affects their lives. The experiences of participants receiving the study medicine will be compared to participants receiving placebo. This will help to understand if PF-08049820 is safe and effective.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet the following criteria:

1. Are 18 years of age or older
2. Have clinical diagnosis of AD for at least 6 months prior to Day 1 and have diagnosis of AD confirmed by photographs
3. Have moderate to severe AD as defined by the following at screening and baseline visits:

   * Affected body surface area (BSA) greater than or equal to 10% and up to 60%;
   * Validated Investigator's Global Assessment (vIGA) greater than or equal to 3;
   * Eczema Area and Severity Index (EASI) greater than or equal to 16;

   AND

   -Peak Pruritis Numeric Rating Scale (PP-NRS) greater than or equal to 4 at screening and a weekly average of greater than or equal to 4 at baseline visit
4. Do not have a suitable prescribed medicine for AD.
5. Body Mass Index (BMI) of 17.5 to 40 kg/m2 and a total body weight greater than 45 kg (100 lbs)

Exclusion Criteria:

Participants must not meet the following criteria:

1. Have an infection that requires treatment
2. Have other skin conditions other than AD
3. Have severe uncontrolled asthma
4. Regular use (more than 2 visits per week) of a tanning booth or phototherapy for AD within 4 weeks of the screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2027-08-23 (Estimated); Study Completion 2027-08-23 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline in Eczema Area and Severity Index (EASI) total score at Week 12 | Week 12

SECONDARY OUTCOMES:
Response based on achieving EASI75 (≥75% improvement from baseline) at scheduled time points | Day 1 through Week 16
Percent change from baseline in EASI total score at scheduled time points other than Week 12 | Day 1 through Week 16
Response based on achieving Validated Investigator's Global Assessment (vIGA) score of clear (0) or almost clear (1) (on a 5-point scale) and a reduction from baseline of >2 points at scheduled time points | Day 1 through Week 16
Response based on achieving ≥4 points of reduction from baseline in weekly averages of Peak Pruritus-Numerical Rating Scale (PP-NRS4) at scheduled time points | Day 1 through Week 16
Incidence of treatment emergent Adverse Events (AEs) and Serious Adverse Events (SAEs), and clinically significant changes in laboratory tests, vital signs and ECGs | Day 1 through Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Clinical Science Institute, Santa Monica, California
  - Gsi Clinical Research, Margate, Florida
  - Skin Research of South Florida, Miami, Florida
  - Goodlettsville Dermatology Research, Goodlettsville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C6231002